CLINICAL TRIAL: NCT04414865
Title: A Prospective, Multi-center, Post-market Registry Study Evaluating Safety and Effectiveness of the Microport™CardioFlow VitaFlow™Transcatheter Aortic Valve System for the Treatment of Severe Aortic Stenosis
Brief Title: VitaFlow™ Transcatheter Aortic Valve System Post-market Study-The LAUNCH Study
Status: Recruiting | Type: Observational
Sponsor: Shanghai MicroPort CardioFlow Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LAUNCH-2020
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single arm, treatment group: Subjects in the treatment group will be implanted with the VitaFlow™ Transcatheter Aortic Valve System
  Interventions: Device: VitaFlow™ Transcatheter Aortic Valve System

INTERVENTIONS:
Device: VitaFlow™ Transcatheter Aortic Valve System — VitaFlow™ Transcatheter Aortic Valve System contains a valve stent-VitaFlow™ Aortic Valve, a delivery system-VitaFlow™ Delivery System,loading tools, a balloon dilatation catheter, and an introducer set

SUMMARY:
The study objective is to evaluate safety and effectiveness/performance of the Microport™ CardioFlow VitaFlow™ Transcatheter Aortic Valve System for the treatment of severe aortic stenosis in the real world settings.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, observational, post-market registry study. The purpose is to evaluate the safety, performance, and effectiveness of the VitaFlow™ Transcatheter Aortic Valve System in the real world settings.Patients will be seen at pre and post procedure, discharge, 30 days, 1 year and annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age≥70 years;
* Symptomatic , calcified, severe, degenerative, native aortic valve stenosis : peak velocity ≥4.0m/s, or mean transvalvular gradient ≥40mmHg(1 mmHg=0.133kPa), or aortic valve area<0.8cm² (or EOA index<0.5cm²/m²);
* The patients considered to be not suitable for surgical aortic valve replacement (SAVR);
* The patient has been informed of the nature of the study, is willing to enroll in the study by signing a patient informed consent and agreeing to the scheduled follow up requirement.

Exclusion Criteria:

* Aortic root anatomy not suitable for the implantation of the transcatheter aortic valve；
* Vascular diseases or anatomical condition preventing the device access；
* Previous implantation of mechanical or bioprosthesis valve in the aortic position；
* Known hypersensitivity or contraindication to all anticoagulation/antiplatelet regimens, to nitinol, contrast media or other relevant elements；
* Ongoing sepsis, including active endocarditis；
* Estimated Life expectancy< 12 months；
* Participating in another trial and the primary endpoint is not achieved.
* Inability to comply with the clinical investigation follow-up or other requirements.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population includes symptomatic patients (≥70 years old ) with calcified, severe, degenerative, native aortic valve stenosis who are not suitable for the surgical aortic valve replacement as assessed by the heart team
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-26 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality at 12 months post implantation | 12 months post implantation
  Rate of all-cause mortality including cardiovascular and non-cardiovascular death

SECONDARY OUTCOMES:
Valve function-mean transvalvular gradient | at discharge, 30 days, 1 year and annually up to 5 years post implantation
  Mean transvalvular gradient measured by transthoracic echocardiography (TTE)(in mmHg)
Valve function-effective orifice area | at discharge, 30 days, 1 year and annually up to 5 years post implantation
  Effective orifice area measured by transthoracic echocardiography (TTE)(in cm^2)
Valve function-degree of prosthetic valve regurgitation | at discharge, 30 days, 1 year and annually up to 5 years post implantation
  Degree of prosthetic valve regurgitation, including paravalvular leak and intravalvular regurgitation measured by transthoracic echocardiography (TTE)
Rate of safety events according to VARC2 | at immediate, 30 days, 1 year and annually up to 5 years post implantation
  Rate of safety events according to VARC2 including all-cause mortality, myocardial infarction, stroke, bleeding, acute kidney injury, vascular complications, new permanent pacemaker implantation
Rate of other TAVI-related complications | at immediate, 30 days, 1 year and annually up to 5 years post implantation
  Rate of other TAVI-related complications including conversion to open surgery, unplanned use of cardiopulmonary bypass, coronary obstruction, ventricular septal perforation, mitral valve apparatus damage or dysfunction, cardiac tamponade, endocarditis, valve thrombosis, valve mal-positioning, TAV-in-TAV, valve related dysfunction requiring repeat procedure (TAVI,SAVR,BAV)
Rate of device success | at immediate post implantation
  Rate of device success, assessed by the access, delivery, deployment and implantation of the device and the prosthetic valve function
Rate of balloon pre-dilatation success | at immediate post implantation
  Rate of balloon pre-dilatation success, assessed by the access, delivery, pre-dilatation and retrieval of the balloon catheter
Rate of balloon post-dilatation success | at immediate post implantation
  Rate of balloon pre-dilatation success, assessed by the access, delivery, post-dilatation and retrieval of the balloon catheter
Rate of procedure success | at immediate post implantation
  Rate of procedure success, assessed by the device success and peri-procedural complications

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ruijing Hospital，Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality